CLINICAL TRIAL: NCT06505785
Title: The Effect of Creative Drama Education on Students' Empathic Tendencies and Emotion Management Skills
Brief Title: The Effect of Creative Drama Education's Effects Tendencies and Emotion Management Skills
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Esra Sayar, Dr, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: AtaturkU-SBF-ES-00
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-07

CONDITIONS: Creative Drama; Emotion Management Skills; Tendencies; Midwifery Student
Keywords: Emotion Management Skills, Tendencies, Creative drama

STUDY DESIGN:
Intervention Model Description: Randomize-control trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The cretive drama group (Experimental): 10 weeks, once a week, each session will last approximately 2 hours and will be facilitated by a trained instructor in creative drama.
  Sessions will include role-playing, improvisation, and scenario-based activities focusing on midwifery care situations, communication with patients, and empathy development.
  Interventions: Other: The creative drama group
- the control group (No Intervention): This group will consist of students who choose another elective course other than the creative drama course, and no interference will be made.

INTERVENTIONS:
Other: The creative drama group — 10 weeks, once a week, each session will last approximately 2 hours and will be facilitated by a trained instructor in creative drama.
  Sessions will include role-playing, improvisation, and scenario-based activities focusing on midwifery care situations, communication with patients, and empathy development.
  Arms: The cretive drama group

SUMMARY:
An experiential and active approach to learning can be implemented in education in higher education through all the arts. In this context, one of the artistic methods that supports active and experiential learning is creative drama. Creative drama is an educational method that is designed to achieve specified cognitive, affective and psychomotor goals and has no age or subject restrictions.This study is planned to examine the effect of the creative drama method on student midwives' empathic tendencies and their ability to manage their emotions.

DETAILED DESCRIPTION:
An experiential and active approach to learning can be applied to higher education through all arts. One of the artistic methods that supports active and experiential learning in this context is creative drama. Creative drama is an educational method designed to impart specific cognitive, affective, and psychomotor objectives, without age or subject limitations. The importance of creative drama lies in its ability to teach through the most realistic experience, by doing and living, thereby enhancing achievement, learning, and retention. Creative drama can be used in midwifery education to bridge the gap between theory and practice, to engage students in group activities where they can explore care practices, events, and relationships, to help students discover knowledge gaps, and to provide deeper learning. It is believed that creative drama supports midwifery students' communication skills , reflective and ethical skills, and critical thinking. Through this method, students can increase their self-awareness, develop empathy by thinking like a patient, and experience the outcomes of midwifery care. Therefore, drama can be used in midwifery education to alleviate fears and anxieties related to clinical birth experiences and to develop empathic skills.

Communication, an essential element of our lives and the foundation of information exchange, plays a significant role in the patient-midwife relationship. Establishing healthy patient-midwife communication, which requires mutual respect, support, and trust, is indispensable for the treatment process. Empathic communication plays a critical role in midwifery, a profession that dates back as far as human existence. Empathy skills, which are crucial in the development of interpersonal communication, enable people to understand the situation of others and socialize with each other.

Birth is both a universal phenomenon and a unique experience. During this process, women need the support of others. Health professionals, especially midwives and obstetricians, have significant responsibilities in providing this support . One of the primary responsibilities of the midwife is to provide emotional and physical support to the woman during labor. To provide this support effectively, midwives need to have well-developed empathy skills. Empathy is the process of accurately understanding another person's feelings and thoughts by putting oneself in their place and communicating this understanding to them.

It is known that emotions are important factors influencing human behavior. Past emotions and the anticipation of future negative events can impact an individual's present. In emotion management, it is important to focus on the present, free from the influence of the past and future.

The management of emotions becomes particularly significant in professions involving a professional identity and human relationships. The healthcare sector is an area where direct and prolonged contact with people occurs, making communication and thus emotion management crucial. Among healthcare professionals, midwives are one of the professions that interact the most with patients or their relatives.

This study aims to examine the effect of the creative drama method on the empathic tendencies and emotion management skills of student midwives.

This research was planned as an experimental type with a pre-test, post-test control group.

Place and Time the Research Was Conducted This study is an experimental study to understand the effectiveness of drama education in developing empathic tendencies and emotion management skills. The research will be conducted experimentally (pretest-posttest design in double groups). Within the 12-week/2-hour training program, drama techniques such as role playing, improvisation, pantomime, making headlines and creating photo frames will be used. The research will be conducted between March 2024 and December 2024 with students who choose the Creative Drama course at Atatürk University Faculty of Health Sciences, Department of Midwifery.

ELIGIBILITY:
Inclusion Criteria:

* No communication problems,
* Conscious,
* Choosing the creative drama course,
* Individuals who volunteer to participate in the study

Exclusion Criteria:

* Communication problems,
* Unconscious,
* No choosing the creative drama course,
* Individuals who no volunteer to participate in the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Midwifery student
Enrollment: 60 (Actual)
Dates: Start 2024-03-30 (Actual); Primary Completion 2024-07-11 (Actual); Study Completion 2024-07-11 (Actual)

PRIMARY OUTCOMES:
Empathic Tendencies | 5-10 minutes
  Empathic Tendency Scale (ETS) was developed by Dökmen (1988) to increase empathy potential in daily life. It is a Likert-type scale and consists of 20 questions and each section is given a score from 1 to 5. 3,6,7,8,11,12,13,15 while adding up the points. Questions
  are collected mutually. The minimum score to be obtained from the scale is 20 and the maximum score is 100. The total score represents the subjects' empathic scores. The higher the score, the higher the empathic feature; The trait of being low indicates that the empathic trait is low. The reliability of the scale is .82.

SECONDARY OUTCOMES:
Emotion Management Skills | 5-10 minutes
  It was developed by Çeçen in 2006. EMS consists of a total of 28 items, 8 of which are positive and 20 are negative. EMS is a 5-point Likert-type self-evaluation performance ranging from Not at All Suitable for Me (1) to Completely Suitable for Me (5). The highest
  score that can be obtained from the scale is 140 and the lowest score is 28. While scoring the scale, reverse scores are converted in cases 1, 3, 4, 5, 6, 7, 9, 11, 13, 14, 15, 16, 18, 20, 22, 23, 24, 25, 27 and 28, which are expressed negatively. . . High scores indicate that individuals are competent in organizing their information. The scale consists of five sub- dimensions; Being able to express emotions verbally 3, 4, 7, 9, 23, 25, 27; Being able to show emotions as they are; 15, 16, 18, 20, 24,28; Ability to control the reactions of negative formations 1, 5, 11, 13; Coping 2, 17, 21, 26; Anger management includes articles 6, 22, and 14.

CONTACTS AND LOCATIONS:
Overall Officials: Faculty Health Science, Study Chair — Ataturk University
Locations (1):
- Ataturk Universty, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No, we don't plan to share individual participant data

REFERENCES:
- [Background] Arveklev SH, Wigert H, Berg L, Burton B, Lepp M. The use and application of drama in nursing education--an integrative review of the literature. Nurse Educ Today. 2015 Jul;35(7):e12-7. doi: 10.1016/j.nedt.2015.02.025. Epub 2015 Mar 21. PMID 25819267
- [Background] Hancer Tok H, Cerit B. The effect of creative drama education on first-year undergraduate nursing student attitudes toward caring for dying patients. Nurse Educ Today. 2021 Feb;97:104696. doi: 10.1016/j.nedt.2020.104696. Epub 2020 Dec 5. PMID 33388550